CLINICAL TRIAL: NCT06300190
Title: Biceps Tenodesis Alone Versus Biceps Tenodesis and Labrum Repair in Superior Labrum Anteroposterior (SLAP) Lesion Type IV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mahrous Fouad Mohamed, Resident of orthopaedic and trauma surgery Assiut university hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Treatment SLAP type IV lesion
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: SLAP Lesion

STUDY DESIGN:
Intervention Model Description: 2 parallel groups selected by Randomisation
Who Masked: Outcomes Assessor
Masking Description: Aim of this study is comparing outcome results of Biceps Tenodesis Alone Versus Biceps Tenodesis and labrum Repair in Superior Labrum Anteroposterior (SLAP) Lesion Type IV
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biceps tenodesis alone (Other)
  Interventions: Procedure: Biceps tenodesis alone
- Biceps tenodesis and repair labrum (Other)
  Interventions: Procedure: Biceps tenodesis and labrum repair

INTERVENTIONS:
Procedure: Biceps tenodesis alone — Biceps tenodesis in superior labrum anteroposterior lesion type IV
  Arms: Biceps tenodesis alone
Procedure: Biceps tenodesis and labrum repair — Biceps tenodesis and labrum repair by anchors in superior labrum anteroposterior lesion type IV
  Arms: Biceps tenodesis and repair labrum

SUMMARY:
Aim of this study is comparing results Biceps Tenodesis Alone Versus Biceps Tenodesis and labrum Repair in Superior Labrum Anteroposterior (SLAP) Lesion Type IV

DETAILED DESCRIPTION:
A SLAP (Superior Labrum Anterior to Posterior) lesion is a specific type of shoulder injury that involves damage to the superior labrum, which is the cartilage rim around the socket of the shoulder joint. This type of injury typically occurs at the long head of the biceps tendon attaches to the labrum. The patient may feel pain, popping sensations and decreased range of motion in the shoulder.1 SLAP lesions are occurring in younger individuals,who playing sports that require repetitive overhead motions and presenting in individuals who have shoulder trauma injury,such as a fall or a direct blow to the shoulder.5There are four main types of SLAP lesions: in this research including Type IV: That is characterized by a bucket-handle tear of the superior labrum that extends into the biceps tendon. The torn portion of the labrum is displaced into the joint and the biceps tendon may be partially or completely detached.The prevalence of SLAP lesions as a cause of shoulder pain is estimated to be around 6-26% in the general population. However, the prevalence can vary depending on the specific population being studied, such as athletes or individuals with specific occupations that involve repetitive overhead activities.Treatment of SLAP type IV is Biceps tenodesis which was recently described, used suture anchor for fixation the biceps tendon to proximal humerus to obtain the stability of glenohumeral muscle. Fixation methods include tenodesis through a bone tunnel, the keyhole method, soft tissue tenodesis to the rotator interval or conjoint tendon, interference screw fixation, and suture anchors tenodesis which have a role in pain relief and maintain biceps muscle strength and have a role in preventing cramping. Recently treatment of SLAP lesion is repairing the labrum using suture anchors with Biceps tenodesis.This study prepared to compare the results of Biceps Tenodesis Alone Versus Biceps Tenodesis and labrum Repair in Superior Labrum Anteroposterior (SLAP) Lesion Type IV ?

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and degenerative etiology.
* No shoulder deformity .
* No inflammatory joint disorders.
* Type of the SLAP is SLAP type IV.

Exclusion Criteria:

* History of the disease.
* Bilateral shoulder.
* DM .
* Epilepsy .
* psychological disturbance.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Clinical outcome by American shoulder elbow score | 12 months
  Examination of the patients and ask them about their pain degree and record the results

REFERENCES:
- See also: American Academy of Orthopaedic Surgeons. (2018). SLAP Tears. Retrieved from https://orthoinfo.aaos.org/en/diseases--conditions/slap-tears/. — http://orthoinfo.aaos.org/en/diseases--conditions/slap-tears/